CLINICAL TRIAL: NCT00950963
Title: Nurse-run, Telephone-based Intervention to Improve Lipids in Diabetics
Brief Title: Nurse Telephone Management of Cholesterol in Diabetes
Acronym: NATCHOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Raymond Estacio, MD, Denver Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 05-509
Record Dates: First submitted 2009-01-12; First posted 2009-08-03 (Estimated); Results first posted 2009-08-03 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: Diabetes, Nurse phone intervention, lipid control
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Counseling; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phone Counseling (Experimental): The telephone outreach intervention was considered an adjunct to usual care. The study nurse focused on optimizing lipids utilizing published guidelines through phone contact.
  Interventions: Behavioral: Phone Counseling
- Standard Care (Active Comparator): Patients in the usual care or control group were contacted at the beginning of the study only if they had not had an LDL level in the previous 12 months. A letter requesting their presentation for an LDL test was sent to their last known address along with a lab slip and a reminder to schedule an appointment with their PCP for follow-up of results. No additional contact was made with them by the study nurses.
  Interventions: Other: Standard Clinical Care

INTERVENTIONS:
Behavioral: Phone Counseling — Patient were contacted on a periodic basis via telephone to address there diabetes care.
  Other Names: Telephone Intervention; Counseling
  Arms: Phone Counseling
Other: Standard Clinical Care — Patients in the usual care or control group were contacted at the beginning of the study only if they had not had an LDL level in the previous 12 months. A letter requesting their presentation for an LDL test was sent to their last known address along with a lab slip and a reminder to schedule an appointment with their PCP for follow-up of results. No additional contact was made with them by the study nurses.
  Other Names: Standard Care
  Arms: Standard Care

SUMMARY:
The current project is evaluating the effect of a nurse-administered phone care in diabetes to improve access to care and healthcare delivery. The setting is a federally qualified community health center serving over 1600 diabetic patients, 80% of whom are Latino. Using our diabetes registry, we have randomly assigned 762 patients to either participate in a telephone-based, nurse-run outreach program (N=381) or to continue with usual care(N=381). Three of our registered nurses learned algorithms addressing management of cholesterol, blood pressure, kidney disease, aspirin use, eye screening, and pneumovax and influenza vaccines. The program began recruitment in September 2005 and has finished follow up in May 2007. The program initially focused only on cholesterol management utilizing national guidelines and algorithms on patients with elevated cholesterol (LDL) levels but has expanded to include glycemic and blood pressure control. We found that Registered Nurses were able and willing to provide telephone care to diabetic patients according to moderately complex algorithms and to track patient data electronically with overall job satisfaction. Overall, the nurses have expressed enthusiasm but have also experience frustrations with maintaining contact and improving motivation in patients. The impact of this program on diabetes outcomes and its cost-effectiveness is currently being analyzed with the goal of implementing this program in our institution.

DETAILED DESCRIPTION:
This randomized, controlled trial tested the effectiveness of a nurse-run, telephone-based intervention to improve lipid control in patients with diabetes. Our patient population is predominantly low-income and Latino. Using our diabetes registry, we randomly assigned 381 patients to continue with their usual care and 381 to participate in our nurse run program. Three registered nurses learned algorithms for diabetes care. These algorithms address management of lipids, glycemic control, blood pressure, nephropathy, aspirin use, eye screening, pneumovax and influenza vaccines, obesity, and cigarette smoking. The nurses were also trained in motivational interviewing techniques and facilitation of patient self-management. The primary goal was to improve lipid control in our diabetic population. Secondary outcomes address blood pressure control, glycemic control, renal function, and medication adherence. In addition, a cost-effective analysis is being performed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients included in Denver Health diabetes registry.
2. Type I and Type II diabetic patients
3. Age >17 years old
4. Actively utilizing Westside Clinic for their primary care (at least two visits in the past year)
5. Speak either English or Spanish.

Exclusion Criteria:We sought to maximize the generalizability of the study and therefore had only minimal exclusion criteria:

1. Pregnant or lactating women
2. Patients with end-stage renal disease (creatinine > 3.0 mg/dl)
3. Patients with a co-morbid illness with life expectancy less than 12 months, (e.g. terminal cancer or Child's Class C hepatic cirrhosis).

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 762 (Actual)
Dates: Start 2005-09; Primary Completion 2007-05 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond O Estacio, MD, Principal Investigator — Denver Health; Henry Fischer, MD, Study Director — Denver Health
Locations (1):
- Denver Health, Westside Clinic, Denver, Colorado, United States

REFERENCES:
- [Background] Fischer H, Mackenzie T, McCullen K, Everhart R, Estacio RO. Design of a nurse-run, telephone-based intervention to improve lipids in diabetics. Contemp Clin Trials. 2008 Sep;29(5):809-16. doi: 10.1016/j.cct.2008.05.011. Epub 2008 Jun 11. PMID 18606250

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of patients began in September 2005 from one community clinic. Study nurses attempted to contact all patients in the control group at the beginning of the study only if they had not had an LDL level in the previous 12 month. An LDL level was obtained to be used as baseline.
Pre-assignment Details: Patients were randomized directly from a registry.
Period: Overall Study
Arm/Group | Phone Counseling | Standard Care
Started | 381 (Patients were randomized from a diabetes registry and were followed as intent to treat) | 381 (Patients were randomized from a diabetes registry and were followed as intent to treat)
Completed | 352 | 357
Not Completed | 29 | 24
Not completed — Lost to Follow-up | 29 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phone Counseling | Standard Care | Total
Number analyzed (Participants) | 381 | 381 | 762
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 252 | 261 | 513
  >=65 years | 129 | 120 | 249
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (12.5) | 58.3 (12.1) | 58.4 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 244 | 218 | 462
  Male | 137 | 163 | 300
Region of Enrollment [Number; unit: participants]
  United States | 381 | 381 | 762

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a Low Density Lipid (LDL) Value Less Than 100 mg/dL
Description: Number of patients with and without cardiovascular disease (CVD) with LDL value less than 100 mg/dL at the end of the study
Time Frame: 18 months
Population: Analysis was per intention to treat.
Measure: Number; unit: Participants
Arm/Group | Phone Counseling | Standard Care
Number analyzed (Participants) | 381 | 381
Participants | 223 | 178

2. Secondary Outcome: Number of CVD Patients With LDL Less Than 70 mg/dL.
Time Frame: 18 months
Population: Analysis was per intention to treat
Measure: Number; unit: Participants
Arm/Group | Phone Counseling | Standard Care
Number analyzed (Participants) | 104 | 102
Participants | 41 | 31

3. Other Pre Specified Outcome: Number of Total Emergency Department (ED) Visits and Hospital Admissions During the Follow up Period.
Description: Evaluate the effect of the intervention on healthcare utilization as defined by ED visits and hospitalizations
Time Frame: 18 months
Population: Analysis per intention to treat
Measure: Number; unit: Number of ED visits and hospitalizations
Arm/Group | Phone Counseling | Standard Care
Number analyzed (Participants) | 381 | 381
Number of ED visits and hospitalizations | 246 | 360

4. Secondary Outcome: Number of Patients With BP Less Than 130/80 mm Hg
Description: Number of patients meeting blood pressure goals as defined by the American Diabetes Association guidelines.
Time Frame: 18 months
Population: Analysis per intention to treat
Measure: Number; unit: participants
Arm/Group | Phone Counseling | Standard Care
Number analyzed (Participants) | 381 | 381
participants | 168 | 191

5. Secondary Outcome: Number of Patients With Hgb A1c Less Than 7 Percent at the End of the Study
Description: Number of patients with Hgb A1c as recommended by the American Diabetes Association guidelines.
Time Frame: 18 months
Measure: Number; unit: Participants
Arm/Group | Phone Counseling | Standard Care
Number analyzed (Participants) | 381 | 381
Participants | 62 | 59

ADVERSE EVENTS:
Time Frame: 5 days
Arm/Group | Phone Counseling | Standard Care
Serious Adverse Events (participants affected / at risk) | 0/381 | 0/381
Other Adverse Events (participants affected / at risk) | 0/381 | 0/381

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No